CLINICAL TRIAL: NCT04516850
Title: An Exploratory Analysis of the Expression of Receptors and Activating Proteases Mediating SARS-CoV-2 Entry and the Association Between HSD3B1 Gene Polymorphisms With Outcomes in SARS-CoV-2 Infected Patients
Brief Title: HSD3B1 Gene Polymorphisms With Outcomes in SARS-CoV-2 Infected Patients
Status: Completed | Type: Observational
Sponsor: Ricardo Pereira Mestre (Other)
Collaborators: Institute of Oncology Research (IOR) (Unknown); Istituto Cantonale di Patologia (Other)
Responsible Party: Sponsor-Investigator, Ricardo Pereira Mestre, MD, Oncology Institute of Southern Switzerland
Organization: Oncology Institute of Southern Switzerland (Other)
Other Study IDs: COVID19-GeneExp
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sub-project 1: nasopharyngeal swabs
  Sub-project 2: tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients tested for COVID-19: The nasopharyngeal swabs taken from patients tested for Covid-19 who resulted infected and non-infected will be analyzed to evaluate the expression of receptors and activating proteases mediating SARS-CoV-2.
  Interventions: Genetic: Expression of receptors and activating proteases
- Patients with mild-moderate and severe SARS-CoV-2 infection: Formalin-fixed paraffin will be analysed to determine the association between polymorphism of the HSD3B1 gene and outcomes in COVID-19 affected patients
  Interventions: Genetic: Polymorphism of the HSD3B1

INTERVENTIONS:
Genetic: Expression of receptors and activating proteases — Level of expression of the mRNA of the genes encoding ACE2, TMPRSS2, TMPRSS4 and AR along with reference genes (beta-actin and EPCAM) in nasopharyngeal swabs taken from patients tested for COVID-19
  Groups: Patients tested for COVID-19
Genetic: Polymorphism of the HSD3B1 — Formalin-fixed paraffin embedded tissue blocks will be amplified using polymerase chain reaction (PCR) based experiments followed by direct sequencing (Sanger sequencing)
  Groups: Patients with mild-moderate and severe SARS-CoV-2 infection

SUMMARY:
The study includes 2 sub-projects.

Sub-project 1: The aim is to evaluate the expression of receptors and activating proteases mediating SARS-CoV-2 entry and spreading in the local population of Ticino.

Sub-project 2: The aim is to investigate the association between the HSD3B1 gene variations and outcome of COVID-19 in the local population of Ticino.

DETAILED DESCRIPTION:
Sub-project 1:

This is an observational retrospective study that aims to evaluate the expression of receptors and activating proteases mediating SARS-CoV-2 entry and spreading in the local population of Ticino. The level of expression of these factors will be compared between infected and non-infected subjects. The sub-project will examine RNA samples from nasopharyngeal swabs taken from subjects tested for COVID-19.

Sub-project 2:

This is a haplotype- and diplotype-based case-control retrospective study that aims to investigate the association between the HSD3B1 gene variations and outcome of COVID-19 in the local population of Ticino. The gene status of HSD3B1 will be defined and compared between two groups of patients: the patients who experienced a severe SARS-CoV-2 infection (severe pulmonary insufficiency, ICU admission, eventually death) and the group with a mild-moderate COVID-19 disease without pulmonary insufficiency and oxygen need.

ELIGIBILITY:
Sub-project 1

Inclusion Criteria:

* Availability of RNA extracted from nasopharyngeal swabs taken from subjects tested for COVID-19;
* Subject is aged 18 years or over;
* Written informed consent (for SARS-CoV-2 positive patients only; see §5 for further details).

Exclusion Criteria:

- Documented refusal.

Sub-project 2

Inclusion Criteria:

* Female and male hospitalized SARS-CoV-2 patients;
* Patient is aged 18 years or over;
* Availability of archival tissue samples collected at any time before SARS-CoV-2 infection for any clinical reason;
* Clinico-pathological characteristics of the COVID-19 and clinical outcomes recorded in the EOC and Clinica Luganese Moncucco database;
* Written informed consent (see §5 for further details).

Exclusion Criteria:

- Documented refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects tested for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Expression of receptors and activating proteases | 1 year
  Determination of the level of expression of the mRNA genes
Prevalencen of olymorphisms of the HSD3B1 | 1 year
  Determination of the prevalence of polymorphisms of the HSD3B1 patients with severe and mild-moderate SARS-CoV-2 infection
Association of polymorphisms of the HSD3B1 | 1 year
  Evaluation of the association of polymorphisms of the HSD3B1 with clinico-pathological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Pereira Mestre, MD, Study Chair — Oncology Institute of Southern Switzerland (IOSI)
Locations (2):
- Switzerland (2):
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona
  - Clinica Luganese Moncucco, Lugano

IPD SHARING:
Plan to Share IPD: No